CLINICAL TRIAL: NCT01359501
Title: Evaluation of the Effects of Chinese Medical Treatment on Leucopenia After Chemotherapy in Breast Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Collaborators: Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government)
Responsible Party: Director of Surgery Department, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DMR99-IRB-259; CCMP99-RD-050 (Other Grant/Funding Number: CCMP99-RD-050)
Record Dates: First submitted 2011-05-01; First posted 2011-05-24 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Leucopenia; Breast Cancer
Keywords: patients receiving chemotherapy
MeSH Terms: conditions — Leukopenia; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chinese medical treatment (Experimental)
  Interventions: Drug: Chinese medical treatment-LCH1
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Chinese medical treatment-LCH1 — Start to take the powder of Chinese herb-LCH1 3g*BID just after the 1st chemotherapy, and Stop 2-3 weeks after the final cycle of chemotherapy.
  Arms: Chinese medical treatment
Drug: Placebo — Start to take the powder of Placebo 3g*BID just after the 1st chemotherapy, and stop 2-3 weeks after the final chemotherapy.
  Arms: Placebo

SUMMARY:
This is a two-year double blind, placebo-controlled, and randomized clinical trial, which is aimed to evaluate the effects of Chinese medical treatment on leucopenia after chemotherapy in breast cancer patients.

DETAILED DESCRIPTION:
The study will be conducted in the Department of Breast Surgery in China Medical University Hospital, Taichung. One hundred newly diagnosed breast cancer patient (age ≧18, Stage I, II, IIIa) will be included. After the diagnosis, the patients will undergo operation. Then, each patient will receive one of the following protocol of chemotherapy according to her pathology report and overall evaluation: "FEC*6", "FEC*4+Taxotere*4", and "FEC*3+Taxotere*3".

Every participator will start to take the powder of Chinese herb-LCH1 after her receiving first time of chemotherapy until she receives the next cycle.(While receiving "FEC", it will be 3 weeks. While receiving "Taxotere", it will be 4 weeks).

Just before receiving the next cycle of chemotherapy, the blood of the participator will be sampled to check her CBC, GOT/GPT, BUN/Cr and tumor maker.

The investigators also adopt the body constitution questionnaire (BCQ) to evaluate the Chinese medical constitutional status, the EORTC QLQ-C30, EORTC QLQ-BR23, and Karnofsky score to evaluate the quality of life, and to evaluate the adverse effects of the adjuvant chemotherapy with the NCI-CTCAE Version 3.0.

Each participator will take the powder of Chinese herb-LCH1 from her first chemotherapy till 3 weeks after the last cycle of chemotherapy. Over all, it will take about 18 weeks (FEC*6) to 28 weeks (FEC*4+Taxotere*4) to complete the treatment.

This study will also investigate the influence of the chemotherapy on the Chinese medical constitutional status, and in order to provide the basis for the complementary treatment for the breast cancer by adjusting and balancing the constitutional status of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed breast cancer patient (age ≧18, Stage I, II, IIIa)
* Receive chemotherapy after operation

Exclusion Criteria:

* Before receiving operation and chemotherapy, the patient already have other chronic diseases.
* Already have hematological malignancy and other lethal disease.
* Pregnant.
* Have severe psychological diseases.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
WBC Count | 21-31 weeks, which depands on the patients' chemotherapy protocol.
  All the patients will be stratified according to her chemotherapy protocol : "FEC*6", "FEC*4+Taxotere*4", and "FEC*3+Taxotere*3".
  The WBC will be checked before receiving each cycle of chemotherapy and at the follow up 3 weeks after the completion of chemotherapy.
  If the participator receives the protocol "FEC*6", her WBC will be checked every 3 weeks for 7 times. It will takes 21 weeks to get the values of WBC at 7 different time point. And it will takes 31 weeks and 24 weeks for participators receive the protocol "FEC*4+Taxotere*4" and "FEC*3+Taxotere*3", respectively.

SECONDARY OUTCOMES:
Score of EORTC QLQ-C30 | 21-31 weeks, which depands on the patients' chemotherapy protocol.
  All the patients will be stratified according to her chemotherapy protocol : "FEC*6", "FEC*4+Taxotere*4", and "FEC*3+Taxotere*3".
  Score of EORTC QLQ-C30 will be evaluated before receiving each cycle of chemotherapy and at the follow up 3 weeks after the completion of chemotherapy.
  If the participator receives the protocol "FEC*6", her score will be checked every 3 weeks for 7 times. It will takes 21 weeks to get the score at 7 different time point. And it will takes 31 weeks and 24 weeks for participators receive the protocol "FEC*4+Taxotere*4" and "FEC*3+Taxotere*3", respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Hwei-Chung Wang, MD., Principal Investigator — Devision of Breast Surgery, China Medical University Hospital; Yi-Chang Su, MD., PhD., Principal Investigator — School of Chinese Medicine, China Medical University
Locations (2):
- Taiwan (2):
  - Devision of Breast Surgery, China Medical University Hospital, Taichung, Taiwan
  - Division of General surgery, Tri-Service General Hospital, Taipei, Taiwan